CLINICAL TRIAL: NCT00641407
Title: Bedtime Insulin Glargine or Bedtime Neutral Protamine Lispro Combined With Sulfonylurea and Metformin in Type 2 Diabetes. A Randomized, Controlled Trial
Brief Title: Bedtime Insulins and Oral Antihyperglycemic Drugs in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Dario Giugliano, MD, PhD, Department of Geriatrics and Metabolic Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGMM-01/2006
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Type 2 Diabetes Mellitus; Hypoglycemia
Keywords: Bedtime insulins; Poorly controlled type 2 diabetes; Glycemic control; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — neutral protamine lispro insulin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: NPL insulin
- 2 (Active Comparator)
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: NPL insulin — Starting dose 10 IU bedtime and then titration
  Arms: 1
Drug: Insulin glargine — 10 IU bedtime and then titration
  Arms: 2

SUMMARY:
The maintenance of nearly normal glycemic levels reduces the risk of diabetic complications, but is difficult to achieve, despite the administration of escalating doses of oral antidiabetic drugs, such as metformin, sulfonylureas, and thiazolidinediones. Most patients eventually require insulin which usually is added when glycemic control with a regimen of oral antidiabetic agents becomes suboptimal.

The aims of the present study were: 1) To compare the clinical efficacy of insulin glargine and neutral protamine lispro (NPL) insulin when added to ongoing oral therapy in poorly controlled type 2 diabetic patients; 2) to find out the possibility to phenotype the patient who may benefit more by the single treatment.

This an open-label, randomized, parallel, 36-week comparative study was performed between January 2007 and March 2008 at a single centre.

DETAILED DESCRIPTION:
Patients were randomized to either NPL (Lilly) or glargine (Lantus, Aventis) to be administered subcutaneously at bedtime. Both insulin formulations consisted of cartridge containing 3 ML of either insulin preparation. Oral antihyperglycemic agents were continued at the prestudy dosages. No dietary advice was given beyond reinforcement of standard guidelines. The initial bedtime insulin dose was 10 IU for all patients with the goal to achieve a target FPG of < 100 mg/dL in both groups. The insulin dose was titrated weekly according to daily self-monitored fasting blood glucose measurements that provide values corresponding closely to laboratory measurements of plasma glucose. The patients were taught to increase their insulin dose by 2 IU if FPG was greater than 100 mg/dL, and by 4 IU if FPG was greater than 180 mg/dL on three consecutive mornings. Before the start of insulin therapy, and at weeks 12, 24 and 36, blood was withdrawn for measurements of full blood counts, electrolytes, creatinine, liver enzymes and lipids. Insulin doses, self-monitored plasma glucose (SMPG), and any events associated with signs or symptoms of hypoglycaemia were recorded in diaries.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 30-70 years, with a duration of known diabetes > 2 years
* And treated with stable doses of two oral antihyperglycemic agents (metformin and sulfonylurea) for at least 90 days were selected for the study
* Body mass index less than 40 kg/m2
* HbA1c level between 7.5 and 10%
* And fasting plasma glucose of 120 mg/dL or greater.

Exclusion Criteria:

* Exclusion criteria included pregnancy or breast-feeding
* Previous use of insulin or other antihyperglycemic drugs
* Investigational drug within the previous 3 months
* Use of agents affecting glycemic control (systemic glucocorticoids, and weight-loss drugs)
* Presence of any clinically relevant somatic or mental diseases
* To minimize the likelihood of including subjects with late-onset type 1 diabetes
* Candidate with a positive test for anti-GAD antibody or with fasting plasma C-peptide less than 0.25 pmol/ml were excluded
* Also excluded were patients with abnormal safety laboratory tests
* Including liver enzymes (ALT, AST, AFOS) higher than three times the upper limit of normal and serum creatinine > 1.4 mg/dL)
* History of drug abuse
* Poor compliance with the 8-point daily glucose profile measurement

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c (HbA1c) level from baseline to end point for each treatment group. | 9 months

SECONDARY OUTCOMES:
Percentage of subjects achieving HbA1c ≤7%, incidence of self-reported hypoglycaemic episodes, comparison of SMPG values from 8-point profiles, insulin doses, and body weight. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Dario Giugliano, MD,PhD, Principal Investigator — Department of Geriatrics and Metabolic Diseases
Locations (1):
- Department of Geriatrics and Metabolic Disease, Naples, Italy

REFERENCES:
- [Background] Yki-Jarvinen H, Kauppinen-Makelin R, Tiikkainen M, Vahatalo M, Virtamo H, Nikkila K, Tulokas T, Hulme S, Hardy K, McNulty S, Hanninen J, Levanen H, Lahdenpera S, Lehtonen R, Ryysy L. Insulin glargine or NPH combined with metformin in type 2 diabetes: the LANMET study. Diabetologia. 2006 Mar;49(3):442-51. doi: 10.1007/s00125-005-0132-0. Epub 2006 Feb 3. PMID 16456680
- [Background] Fritsche A, Schweitzer MA, Haring HU; 4001 Study Group. Glimepiride combined with morning insulin glargine, bedtime neutral protamine hagedorn insulin, or bedtime insulin glargine in patients with type 2 diabetes. A randomized, controlled trial. Ann Intern Med. 2003 Jun 17;138(12):952-9. doi: 10.7326/0003-4819-138-12-200306170-00006. PMID 12809451
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B. Management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: update regarding thiazolidinediones: a consensus statement from the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2008 Jan;31(1):173-5. doi: 10.2337/dc08-9016. No abstract available. PMID 18165348